CLINICAL TRIAL: NCT06152887
Title: Treatment of Pain and Sensory Dysfunction in Diabetic Neuropathy by Brain Neuromodulation
Brief Title: Noninvasive Cortical Neurostimulation For Diabetic Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jens Brøndum Frøkjær (Other)
Collaborators: Novo Nordisk A/S (Industry); Vissing fonden (Unknown)
Responsible Party: Sponsor-Investigator, Jens Brøndum Frøkjær, Principal Investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NOPAIN study
Record Dates: First submitted 2023-08-28; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Neuropathy, Painful; Diabetes Mellitus, Type 1
Keywords: tDCS treatment; noninvasive cortical stimulation
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus, Type 1 | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCs (Active Comparator): Active tDCS will be administered through a pair of conductive rubber electrodes covered by saline soaked sponges (35 cm2). The current will be delivered continuously at 2 mA for 30 min through a battery-driven constant-current stimulator. An anodal electrode is placed above the primary motor cortex, M1, while a cathode is placed above the contralateral supraorbital area.
  Interventions: Device: Sooma Oy (tDCS), Helsinki, Finland
- Sham tDCS (Sham Comparator): Sham stimulation will be delivered to the motor cortex using a sham tDCS device that delivers a direct current for 30 seconds at the beginning and end of tDCS to provide sensory experiences similar to active stimulation.
  Interventions: Device: Sooma Oy (Sham), Helsinki, Finland

INTERVENTIONS:
Device: Sooma Oy (tDCS), Helsinki, Finland — Using the 2-channel neuro-stimulator Sooma tDCS equipment we provide 20 minutes of 2 mA anodal stimulation of the primary motor cortex (M1)
  Arms: Active tDCs
Device: Sooma Oy (Sham), Helsinki, Finland — For the sham treatment, an electrical current will also be increased from 0 mA to 2 mA over the first 30 seconds, however, the current will be ramped back down to 0 mA after the initial ramp-up phase and no stimulation is delivered for the rest of the treatment.
  Arms: Sham tDCS

SUMMARY:
To investigate whether transcranial direct current stimulation can alleviate pain and sensory related disturbances in individuals with type 1 diabetes and peripheral neuropathy through neuromodulation of the CNS as compared to sham treatment.

DETAILED DESCRIPTION:
This study is a randomized, cross-over, controlled investigation. The overall objective of this study is to assess the pain-relieving effect of four weeks' transcranial direct current stimulation (tDCS) in individuals with type 1 diabetes and painful polyneuropathy not responding adequately to traditional pharmacological pain treatment, in comparison to the effect of four weeks' sham treatment. Both treatments will be performed using a commercially available and validated device called Sooma tDCS. Sooma tDCS device is a non-invasive neurostimulator that has been CE-marked for the treatment of depression, chronic pain including neuropathic pain and fibromyalgia. The study will begin with a 2-week baseline registration period, in which the patients will receive no treatment. Next, the baseline period will be followed by a 4-week treatment period where the subjects will be randomized to either active treatment or sham treatment. Afterwards, a wash-out period of 6 weeks will occur. Finally, in the second treatment period the patients will switch in treatment assignment, meaning that patient who received active treatment will now receive sham treatment and vice versa. During both treatments, the patients will be asked to self-administer one stimulation dose daily, five times a week. During the whole study, subjects will be asked to complete a pain diary and several questionnaires. Moreover, at the beginning and end of each treatment period (four times), all subjects will undergo testing which will include brain magnetic resonance imaging (MRI) and quantitative sensory testing (QST). The primary efficacy parameters to be evaluated are short and longer lasting alleviation of clinical chronic pain and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years.
* Type-1 diabetes
* Clinically established peripheral neuropathy
* DN4 of ≥4 points indicating that the patient is suffering from neuropathic pain.
* NRS pain scores >3
* Acceptable screening blood samples according to medical judgement
* Signed informed consent

Exclusion Criteria:

* Contraindications to MRI
* Not being able to understand Danish (written and/or verbally)
* Not being able to comply with the study procedures including home-treatment e.g., due to senile dementia, etc.
* Previous brain surgery
* Present alcohol or drug abuse
* Major mental and psychiatric disorders
* Pregnancy
* Active cancer-disease
* Known neural damage or disease in the neural system (e.g., MS or Guillain-Barre) other than diabetic neuropathy
* Previous chemotherapy or intake of experimental medicine
* Active herpes simplex virus or varicella zoster virus infection or known HIV
* Other reasons for limb pain (e.g., critical limb ischemia and lower back pain with radiating pain etc.)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in numeric rating scale (NRS) scores in pain diary | 20 weeks
  The primary clinical efficacy parameter to be evaluated is pain relief. In the clinical part of the study the efficacy is assessed as changes in the daily experience of pain, which will be measured using a patient pain diary based on the NRS. Maximum intensity and average daily NRS will be recorded on daily basis.
  Minimum: 0 Maximum: 10

SECONDARY OUTCOMES:
Brief Pain Inventory questionnaire (mBPI) | Baseline, week 4 (treatment I), week 10, week 14 (treatment II), week 18 (follow-up).
Neuropathy Total Symptom Score-6 (NTSS-6) | Baseline, week 4 (treatment I), week 10, week 14 (treatment II), week 18 (follow-up).
  A score >0 indicates the presence of >1 sensory symptom. Clinically significant symptoms are defined as an NTSS-6 total score >6 points.
Hospital Anxiety and Depression Scale (HADS) | Baseline, week 4 (treatment I), week 10, week 14 (treatment II), week 18 (follow-up).
  HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
Brain MRI | Baseline, week 4 (treatment I), week 10, week 14 (treatment II), week 18 (follow-up).
  Resting state functional MRI will be employed to detect brain activity and functional connectivity changes based on BOLD signals before and after treatment of each patient.
Quantitative sensory testing | Baseline, week 4 (treatment I), week 10, week 14 (treatment II), week 18 (follow-up).
  QST includes temporal summation, pressure pain thresholds, and conditioned pain modulation (CPM).

CONTACTS AND LOCATIONS:
Overall Officials: Jens Brøndum Frøkjær, MD, Ph.D, Principal Investigator — Professor and Chief Physician at Aalborg University Hospital, Department of Radiology
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark